CLINICAL TRIAL: NCT00165464
Title: A Phase II Trial of Taxotere, Cisplatin, and Irinotecan in Advanced Esophageal and Gastric Cancer
Brief Title: Taxotere, Cisplatin and Irinotecan (CPT-11) for Esophagogastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Aventis Pharmaceuticals (Industry)
Responsible Party: Peter C. Enzinger, MD, Dana-Farber Cancer Institute/Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-140
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Esophageal Cancer; Gastric Cancer; GE Junction Cancer
Keywords: Esophageal Cancer; Gastric Cancer; GE Junction; Cisplatin; Taxotere; CPT-11; Irinotecan
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Docetaxel; Cisplatin; Irinotecan

INTERVENTIONS:
Drug: Taxotere — Given once weekly for 2 weeks followed by a one week rest period (1 cycle is 3 weeks) Participants may continue on treatment unless there is disease progression or intolerable toxicities.
Drug: Cisplatin — Given once weekly for 2 weeks followed by a one week rest period (1 cycle is 3 weeks) Participants may continue on treatment unless there is disease progression or intolerable toxicities.
Drug: Irinotecan — Given once weekly for 2 weeks followed by a one week rest period (1 cycle is 3 weeks) Participants may continue on treatment unless there is disease progression or intolerable toxicities.

SUMMARY:
This is a phase II study of taxotere, cisplatin and irinotecan (CPT-11) used in combination to treat metastatic esophageal and gastric cancer in an effort to see what effects (good and bad) the combination may have on the patients cancer.

DETAILED DESCRIPTION:
* Taxotere, cisplatin and irinotecan will be administered to the patient once weekly for 2 weeks followed by a one week rest period (1 cycle is 3 weeks).
* Patients will also receive corticosteroids, intravenous hydration and anti-emetic therapy prior to each treatment.
* A physical exam and bloodwork will be done each week of the treatment and every 2 cycles, reassessment of the tumor by the same imaging method to determine the baseline size will be conducted.
* Patients will remain on the study unless disease progression or intolerable toxicity occur.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, incurable esophageal or gastric carcinoma (carcinoma = adenocarcinoma or squamous cell carcinoma)
* Measurable disease > 1cm (longest diameter) by spiral CT scan or > 2cm by other radiographic technique.
* Lesions must be measurable in at least one dimension.
* Bone lesions, ascites and effusions are not measurable.
* Irradiated lesions are not measurable yet lesions arising in previously irradiated fields are measurable.
* Age 18+ years.
* ECOG performance status 0 or 1.
* Life expectancy greater than 12 weeks.
* Adequate bone marrow function.
* Adequate renal function: creatinine equal to or less than 1.5 mg/dl.
* SGOT less than 2.5 x institutional upper limit of normal if alkaline phosphatase is within institutional upper limit of normal.
* Alkaline phosphatase less than 4.0 x upper limit of normal if SGOT is within institutional upper limit of normal.
* For patients with both SGOT and alkaline phosphatase elevations, SGOT must be less than 1.5 x institutional upper limit of normal and alkaline phosphatase must be less 2.5 x institutional upper limit of normal. For patients with liver metastases, however, SGOT may be < 3.0 x institutional upper limit of normal and alkaline phosphatase may be < 5.0 x institutional upper limit of normal as long as the total bilirubin is within the institutional upper limit of normal.

Exclusion Criteria:

* No prior chemotherapy (except as part of pre- or post-operative therapy, completed > 1 year prior to start date of this protocol).
* Patients who have received prior pelvic radiation therapy are ineligible. Other prior radiation therapy, however, is permitted, provided at least 4 weeks have elapsed since completion of this therapy and the initiation of this protocol.
* No myocardial infarction in the past six months.
* No major surgery in the past three weeks.
* No uncontrolled serious medical or psychiatric illness.
* No uncontrolled diarrhea.
* Patients with a peripheral neuropathy > grade 1 will be excluded.
* Women of childbearing potential must have a negative pregnancy test. Men and women of childbearing potential must use adequate contraception.
* No clinically apparent central nervous system metastases or carcinomatous meningitis.
* No other active malignancy other than non-melanoma skin cancer or in-situ cervical carcinoma. A resected cancer (other than in-situ carcinoma) must have demonstrated no evidence of recurrence for at least 3 years.
* Patients with history of severe hypersensitivity to irinotecan, cisplatin, taxotere or drugs formulated with polysorbate 80 must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-08; Primary Completion 2005-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the response rate of patients with esophageal or gastric carcinoma to weekly Taxotere, Cisplatin, and Irinotecan (CPT-11).

SECONDARY OUTCOMES:
To assess the duration of response and overall survival of patients with esophageal or gastric carcinoma to weekly Taxotere, Cisplatin, and Irinotecan.
To assess the toxicity of this combination in esophageal or gastric carcinoma. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Enzinger PC, Ryan DP, Clark JW, Muzikansky A, Earle CC, Kulke MH, Meyerhardt JA, Blaszkowsky LS, Zhu AX, Fidias P, Vincitore MM, Mayer RJ, Fuchs CS. Weekly docetaxel, cisplatin, and irinotecan (TPC): results of a multicenter phase II trial in patients with metastatic esophagogastric cancer. Ann Oncol. 2009 Mar;20(3):475-80. doi: 10.1093/annonc/mdn658. Epub 2009 Jan 12. PMID 19139178